CLINICAL TRIAL: NCT06589934
Title: Clinical Study of CT 5400 RT for Precise Image Validation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Clinical & Medical Affairs Global (Industry)
Collaborators: Philips Healthcare (Suzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 300079
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Precise Image (AI Reconstruction Feature of CT 5400 RT System)

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes

ARMS (1):
- Image quality (Experimental): Diagnostic Test -Good and excellent rate of PI image quality is greater than or equal to 95%. PI image quality will be assessed by using the retrospective image raw data obtained from CT 5400 RT (applicable body parts include: head, neck, chest, abdomen and coronary)
  Interventions: Diagnostic Test: Precise Image

INTERVENTIONS:
Diagnostic Test: Precise Image — Image reconstruction software

SUMMARY:
The purpose of this study is to evaluate the effectiveness of the Precise Image (PI), an AI feature of CT 5400 RT System

ELIGIBILITY:
Inclusion Criteria:

* 30 image raw data generated from CT 5400 RT system validation clinical trial (protocol name: Clinical study of CT 5400 RT for system validation, ClinicalTrials.gov ID: NCT06466577)
* Applicable body parts include: head, neck, chest, abdomen and coronary

Exclusion Criteria:

* Raw data is considered inappropriate for inclusion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2025-01-25 (Actual); Primary Completion 2025-01-25 (Actual); Study Completion 2025-03-25 (Actual)

PRIMARY OUTCOMES:
Clinical image quality(IQ) | 14 days (anticipated)
  Image quality will be assessed by Likert score (1-5)

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Public Health Clinical Center, Shanghai, Shanghai Municipality, China